CLINICAL TRIAL: NCT05131204
Title: A Randomized, Open-Label, Eculizumab and Ravulizumab Controlled Study to Evaluate the Efficacy and Safety of Pozelimab and Cemdisiran Combination Therapy in Patients With Paroxysmal Nocturnal Hemoglobinuria Who Are Currently Treated With Eculizumab or Ravulizumab
Brief Title: Efficacy and Safety of the Combination of Pozelimab and Cemdisiran Versus Continued Eculizumab or Ravulizumab Treatment in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria
Acronym: ACCESS 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision not related to efficacy or safety.
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R3918-PNH-2022; 2020-002761-33 (EudraCT Number)
Record Dates: First submitted 2021-11-12; First posted 2021-11-23 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab; ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pozelimab and Cemdisiran (Experimental): Randomized 1:1
  Interventions: Drug: Cemdisiran; Drug: Eculizumab; Drug: Pozelimab; Drug: Ravulizumab
- Anti-C5 standard-of-care (Experimental): Randomized 1:1
  Interventions: Drug: Eculizumab; Drug: Ravulizumab

INTERVENTIONS:
Drug: Cemdisiran — Administered per protocol
  Other Names: ALN-CC5
  Arms: Pozelimab and Cemdisiran
Drug: Eculizumab — Administered per protocol
  Other Names: Soliris
Drug: Pozelimab — Administered per protocol
  Other Names: REGN3918
  Arms: Pozelimab and Cemdisiran
Drug: Ravulizumab — Administered per protocol
  Other Names: ALXN1210; Ultomiris

SUMMARY:
The primary objective of the study is:

To evaluate the effect of pozelimab and cemdisiran combination therapy on hemolysis, as assessed by lactate dehydrogenase (LDH), after 36 weeks of treatment, in patients with PNH who switch from eculizumab or ravulizumab therapy versus patients who continue their eculizumab or ravulizumab therapy

The secondary objectives of the study are to:

* Evaluate the effect of pozelimab and cemdisiran combination treatment versus anti-C5 standard-of-care treatment (eculizumab or ravulizumab) on the following:

  * Transfusion requirements and transfusion parameters
  * Measures of hemolysis: LDH control, breakthrough hemolysis, and inhibition of CH50
  * Hemoglobin levels
  * Fatigue as assessed by Clinical Outcome Assessments (COAs)
  * Health-related quality of life (HRQoL) as assessed by COAs
  * Safety and tolerability
* To assess the concentrations of total pozelimab and either total eculizumab or total ravulizumab in serum and total cemdisiran and total C5 protein in plasma
* To assess the immunogenicity of pozelimab and cemdisiran

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of PNH confirmed by a history of high-sensitivity flow cytometry from prior testing
2. Treated with eculizumab or ravulizumab prior to screening visit as described in the protocol Note: Biosimilars are not permitted, unless approved by the Sponsor

Key Exclusion Criteria:

1. Patients with a screening LDH >1.5 × ULN who have not taken their C5 inhibitor within the labeled dose interval at the dose prior to the screening LDH assessment
2. Receipt of an organ transplant, history of bone marrow transplantation or other hematologic transplant
3. Body weight < 40 kilograms at screening visit
4. Any use of complement inhibitor therapy other than eculizumab or ravulizumab in the 26 weeks prior to the screening visit or planned use during the study with the exception of study treatments
5. Not meeting meningococcal vaccination requirements for eculizumab or ravulizumab according to the current local prescribing information (where available) and at a minimum documentation of meningococcal vaccination within 5 years prior to screening visit.
6. Any contraindication for receiving Neisseria meningitidis vaccination.
7. Positive for hepatitis B, and/ or hepatitis C as described in the protocol
8. History of cancer within the past 5 years, except for adequately treated basal cell skin cancer, squamous cell skin cancer, or in situ cervical cancer
9. Participation in another interventional clinical study (except R3918-PNH-2021) or use of any experimental therapy within 30 days before screening visit or within 5 half-lives of that investigational product, whichever is greater, with the exception of eculizumab or ravulizumab.
10. Patients with functional or anatomic asplenia

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Research Facility, Whittier, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 140 participants were expected to be enrolled, however, due to feasibility: five participants were screened and 3 were randomized and treated. There were 2 screen failures.
Period: Overall Study
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Sponsor request | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  Asian | 1 | 1 | 2
  American Indian or Alaska Native | 0 | 0 | 0
  Other | 0 | 0 | 0
  Unknown | 0 | 0 | 0
  Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Lactate Dehydrogenase (LDH) From Baseline to Week 36
Time Frame: From baseline to week 36
Population: Due to Early Termination, this endpoint was removed from the Statistical Analysis Plan and data was not collected for primary and secondary endpoints.
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Transfusion Avoidance After Day 1 Through Week 36
Description: Participants who do not receive a red blood cell (RBC) transfusion as per protocol algorithm based on post baseline hemoglobin values
Time Frame: Day 1 through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With Transfusion Avoidance From Week 4 Through Week 36
Description: Participants who do not receive an RBC transfusion as per protocol algorithm based on post baseline hemoglobin values
Time Frame: Week 4 through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Breakthrough Hemolysis After Day 1 Through Week 36
Description: Participants with an increase in LDH with concomitant signs or symptoms associated with hemolysis as described in the protocol
Time Frame: Day 1 through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Breakthrough Hemolysis From Week 4 Through Week 36
Description: as for outcome 4
Time Frame: Week 4 (day 29) through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With Hemoglobin Stabilization After Day 1 Through Week 36
Description: Participants who do not receive an RBC transfusion and have no decrease in hemoglobin level as defined in the protocol
Time Frame: Day 1 through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants With Hemoglobin Stabilization From Week 4 Through Week 36
Description: Participants who do not receive an RBC transfusion and have no decrease in hemoglobin level as defined in the protocol
Time Frame: Week 4 (day 29) through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Participants With Adequate Control of LDH From Week 8 Through Week 36
Description: Percentage of participants with adequate control of LDH as defined in the protocol
Time Frame: Week 8 (day 57) through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Participants With Adequate Control of LDH After Day 1 Though Week 36
Description: Percentage of participants with adequate control of LDH as defined in the protocol
Time Frame: Day 1 through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percentage of Participants Who Maintained Adequate Control of Hemolysis From Week 8 Through Week 36
Description: Percentage of participants with adequate control of LDH as defined in the protocol
Time Frame: Week 8 through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percentage of Participants Who Maintained Adequate Control of Hemolysis After Day 1 Through Week 36
Description: Percentage of participants with adequate control of LDH as defined in the protocol
Time Frame: Day 1 through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Participants With Normalization of LDH From Week 8 Through Week 36
Description: Percentage of participants with normalization of LDH as defined in the protocol
Time Frame: Week 8 (day 57) through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Percentage of Participants With Normalization of LDH After Day 1 Through Week 36
Description: Percentage of participants with normalization of LDH as defined in the protocol
Time Frame: Day 1 through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Fatigue as Measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Scale From Baseline to Week 36
Description: The FACIT-Fatigue is a 13 item, self-administered clinical outcome assessment (COA) assessing an individual's level of fatigue during their usual daily activities over the past week. This questionnaire is part of the FACIT measurement system, a compilation of questions measuring health related quality of life (QoL) in patients with cancer and other chronic illnesses. The FACIT-Fatigue assesses the level of fatigue using a Likert scale ranging from 0 (not at all) to 4 (very much). Scores range from 0 to 52, with higher scores indicating greater fatigue.
Time Frame: From baseline to week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change in Physical Function (PF) Score on the European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 Items (EORTC-QLQ-C30) From Baseline to Week 36
Description: EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including global health status/quality of life, functional Scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
Time Frame: From baseline to week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change in Global Health Status (GHS)/QoL Scale Score on the EORTC-QLQ-C30 From Baseline to Week 36
Description: EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including global health status/quality of life, functional Scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea and vomiting, and pain), and 7 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, sleep and financial difficulties). Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
Time Frame: From baseline to week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Rate of RBCs Transfused Per Protocol Algorithm After Day 1 Through Week 36
Description: Per protocol algorithm
Time Frame: Day 1 through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Rate of RBCs Transfused Per Protocol Algorithm From Week 4 Through Week 36
Description: Per protocol algorithm
Time Frame: Week 4 through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Number of Units of RBCs Transfused Per Protocol Algorithm After Day 1 Through Week 36
Description: Per protocol algorithm
Time Frame: Day 1 through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number of Units of RBCs Transfused Per Protocol Algorithm From Week 4 Through Week 36
Description: Per protocol algorithm
Time Frame: Week 4 through week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Change in Hemoglobin Levels From Baseline to Week 36
Description: Per protocol algorithm
Time Frame: From baseline to week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Incidence of Treatment Emergent Serious Adverse Events (SAEs)
Description: Treatment period and safety follow up period
Time Frame: Up to week 29
Measure: Number; unit: Events
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 2 | 1
Events | 0 | 0

23. Secondary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs) of Special Interest
Description: Treatment period and safety follow up period
Time Frame: Up to week 29
Measure: Number; unit: Events
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 2 | 1
Events | 1 | 0

24. Secondary Outcome: Incidence of TEAEs Leading to Treatment Discontinuation
Description: Treatment period and safety follow up period
Time Frame: Up to week 29
Measure: Number; unit: Events
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 2 | 1
Events | 0 | 0

25. Secondary Outcome: Change in Total CH50 From Baseline to Week 36
Time Frame: From baseline to week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Percent Change in Total CH50 From Baseline to Week 36
Time Frame: From baseline to week 36
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Concentration of Total C5 in Plasma Through Week 62
Description: Treatment period and safety follow up period
Time Frame: Through week 62
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Concentrations of Total Pozelimab in Serum Through Week 62
Description: Treatment period and safety follow up period
Time Frame: Through week 62
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Concentrations of Total Cemdisiran in Plasma Through Week 32
Description: Treatment period
Time Frame: Through week 32
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Concentrations of Total Eculizumab in Serum Through Week 40
Description: Treatment period
Time Frame: Through week 40
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Concentrations of Total Ravulizumab in Plasma Through Week 44
Description: Treatment period
Time Frame: Through week 44
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Incidence of Treatment Emergent Anti-drug Antibodies (ADAs) to Pozelimab Through Week 62
Description: Treatment period and safety follow up period
Time Frame: Through week 62
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Incidence of Treatment Emergent ADAs to Cemdisiran Through Week 62
Description: Treatment period and safety follow up period
Time Frame: Through week 62
Population: as for outcome 1
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to week 29
Arm/Group | Pozelimab and Cemdisiran | Anti-C5 Standard-of-care
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pozelimab and Cemdisiran (N=2) | Anti-C5 Standard-of-care (N=1)
Injection site rash (General disorders) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
20Dec2022 - Due to feasibility challenges related to enrollment and not due to efficacy or safety concerns, the sponsor terminated the study early and discontinued participant enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT05131204/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT05131204/SAP_001.pdf